CLINICAL TRIAL: NCT00943384
Title: Prospective, Multi-Center Clinical Outcomes Study Evaluating the chronOS Strip Combined With Bone Marrow Aspirate Plus Local Bone for Posterolateral Lumbar Interbody Fusion or Lumbosacral Interbody Fusion
Brief Title: Prospective, Multi-Center Clinical Outcomes Study Evaluating the chronOS Strip Combined With Bone Marrow Aspirate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: chronOS-050709
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Degeneration of Lumbar Intervertebral Disc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chronOS Strip (Experimental): This is a single arm, outcome study for treatment of patients with degenerative disc disease (DDD), with or without stenosis, with interbody fusion, posterolateral pedicle screw system, and the study device (chronOS Strip).
  Interventions: Device: chronOS Strip

INTERVENTIONS:
Device: chronOS Strip — chronOS strip combined with bone marrow aspirate plus local bone
  Other Names: beta-tricalcium phosphate

SUMMARY:
The chronOS Strip is a synthetic bone void filler manufactured from chronOS beta-tricalcium phosphate (β-TCP) granules and a resorbable polymer [poly(lactide co-ε-caprolactone)]. The chronOS Strip, combined with autogenous bone and/or bone marrow or autograft, is intended to be used in the spine for posterolateral fusion.

The purpose of this prospective, multi-center clinical case series was to evaluate posterolateral fusion rates in a prospective series of patients with degenerative disc disease. The surgical procedure consisted of instrumented posterolateral fusion with interbody support. The chronOS Strip, combined with bone marrow aspirate and local bone, was applied to the posterolateral gutters.

ELIGIBILITY:
Inclusion Criteria:

1. Has the following indication for posterolateral fusion (transverse process and facet fusion) with posterior rod and screw fixation:

   • Degenerative Disc Disease (DDD), with or without stenosis. Diagnosis of DDD requires back and/or leg (radicular) pain along with:
   1. Instability (≥ 3 mm translation or ≥ 5° angulation); or
   2. MRI confirmation of Modic Type 1 or Type 2 changes; or
   3. High intensity zones in the disc space.
2. Has one or two motion segment(s) to be fused between L2 and S1;
3. Skeletally mature adult, at least 18 years of age at the time of surgery;
4. Oswestry Low Back Pain Disability Questionnaire score ≥ 30 (out of 100);
5. Has completed at least 6 months of conservative therapy, which may include physical therapy, bracing, systemic or injected medications;
6. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to scheduled visits, treatment plan, completing forms, and other study procedures;
7. Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Three or more motion segments to be fused;
2. Degenerative scoliosis, defined as Cobb angle > 10° at any level in lumbar spine;
3. Has had a previous interbody fusion or posterolateral fusion attempt at any level of the lumbar spine;
4. Active systemic or local infection;
5. Known or documented history of communicable disease, including AIDS and HIV;
6. Active Hepatitis (receiving medical treatment within two years);
7. Active rheumatoid arthritis, non-controlled diabetes mellitus, or any other medical condition(s) that would represent a significant increase in surgical risk or interfere with normal healing;
8. Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months;
9. Known history of Paget's disease, osteomalacia, or any other metabolic bone disease;
10. Osteopenia or Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a dual energy x-ray absorptiometry (DXA) bone mineral density measurement. If DXA is required, exclusion will be defined as a DXA bone density measured T score less than or equal to -1.0.
11. Morbid obesity defined as a body mass index > 40 kg/m2 or weight more than 100 pounds over ideal body weight;
12. Active malignancy. A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy for more than 5 years;
13. Current or recent history (within last 2 years) of substance abuse (e.g., recreational drugs, narcotics, or alcohol);
14. Pregnant or planning to become pregnant during study period;
15. Involved in study of another investigational product that may affect outcome;
16. History of psychosocial disorders that could prevent accurate completion of self reporting assessment scales;
17. Patients who are incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hartford Hospital, Hartford, Connecticut
  - Bay Area Neurosurgery, Brandon, Florida
  - Atlanta Neurosurgical Associates, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Boston Spine Group, Newton, Massachusetts
  - Southern New York Neurosurgical Group, Johnson City, New York
  - The Rothman Institute, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Dept. of Neurosurgery, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center Department of Neurosurgery/Spine Research, Nashville, Tennessee
  - Orthopaedic and Spine Center, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- chronOS Strip: Patients with DDD (with or without stenosis) were treated at one or two contiguous levels between L1 and S1 (inclusive) with interbody fusion and a posterolateral pedicle screw system. The study device (chronOS Strip) was applied to the posterolateral gutters combined with bone marrow aspirate and local bone.
Period: Overall Study
Arm/Group | chronOS Strip
Started | 104 (104 subjects consented and underwent additional screening to determine eligibility to participate)
Treated | 81 (81 subjects were eligible and willing to participate in the study and were treated)
Treated on Protocol | 76 (5 subjects were treated off protocol due to intraoperative decisions made by the surgeon)
Completed | 55 (evaluated at the Month 24 visit with complete or partial data)
Not Completed | 49
Not completed — Dispositioned prior to treatment | 23
Not completed — Treated off protocol-protocol violation | 5
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Number of subjects treated per protocol
Arm/Group | chronOS Strip
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 36
Level(s) treated [Number; unit: participants] — Subjects were treated at one or two contiguous levels from L2 through S1
  participants
    One-level, L2-3 | 1
    One-level, L3-4 | 1
    One level, L4-5 | 22
    One-level, L5-S1 | 18
    Two-level, L3-5 | 8
    Two-level, L4-S1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Posterolateral Fusion Success
Description: The primary outcome for posterolateral fusion status was a composite endpoint incorporating posterior bridging bone status, intersegmental motion (angular and translational motion) and posterior hardware status. To have successful posterolateral fusion, a subject had to be successful in all four components at all levels under investigation. Failure to meet any one of the four components indicated failed posterolateral fusion status.
Time Frame: Month 24
Population: The primary endpoint was evaluated for the per-protocol population. Of the 55 patients who were evaluated at the Month 24 visit, six patients were missing complete radiographic data needed to evaluate the primary endpoint.
Measure: Number; unit: participants
Arm/Group | chronOS Strip
Number analyzed (Participants) | 49
participants | 45

2. Secondary Outcome: Oswestry Disability Index (ODI)
Description: The Oswestry Low Back Pain Disability Questionnaire was self-administered to each subject preoperatively and at each clinical follow up examination. Each of the ten questions had six ordered responses coded on a scale from zero to five. The scale ranges from 0-100. A higher score indicates a higher level of disability, and a negative percent change (post surgery minus baseline) indicates improved function.
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
units on a scale | 20.3 (17.5)

3. Secondary Outcome: Percent Change in Oswestry Disability Index (ODI)
Description: The Oswestry Low Back Pain Disability Questionnaire was self-administered to each subject preoperatively and at each clinical follow up examination. Each of the ten questions had six ordered responses coded on a scale from zero to five. The scale ranges from 0-100. A higher score indicates a higher level of disability, and a negative percent change (post surgery minus baseline) indicates improved function. Percent change in ODI score was calculated as: [(Month 24-Baseline)/Baseline]*100%.
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
percent change | -61.6 (28.7)

4. Secondary Outcome: Back Pain on Visual Analog Scale
Description: The subjects completed questionnaires assessing the intensity of pain experienced in the back at the preoperative visit and at all visits postoperatively. Pain intensity was rated on a scale where zero indicated no pain, and 100 represented the worst possible pain.
Time Frame: Month 24
Population: Of the 55 subjects who were evaluated at Month 24, two were missing back pain data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Strip
Number analyzed (Participants) | 53
units on a scale | 29.5 (27.3)

5. Secondary Outcome: Percent Change in Back Pain on Visual Analog Scale
Description: The subjects completed questionnaires assessing the intensity of pain experienced in the back at the preoperative visit and at all visits postoperatively. Pain intensity was rated on a scale where zero indicated no pain, and 100 represented the worst possible pain. A negative change (post surgery minus baseline) indicated an improvement. Percent change was calculated as: [(Month 24-Baseline)/Baseline]*100%.
Time Frame: Month 24
Population: Back pain was assessed in the per-protocol population. Of the 55 subjects who were evaluated at the Month 24 visit, two were missing data related to back pain.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | chronOS Strip
Number analyzed (Participants) | 53
percent change | -56.6 (52.8)

6. Secondary Outcome: Leg Pain on Visual Analog Scale
Description: The subjects completed questionnaires assessing the intensity of pain experienced in the leg at the preoperative visit and at all visits postoperatively. Pain intensity was rated on a scale where zero indicated no pain, and 100 represented the worst possible pain.
Time Frame: Month 24
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
units on a scale | 21.1 (28.1)

7. Secondary Outcome: Percent Change in Leg Pain on Visual Analog Scale
Description: The subjects completed questionnaires assessing the intensity of pain experienced in the leg at the preoperative visit and at all visits postoperatively. Pain intensity was rated on a scale where zero indicated no pain, and 100 represented the worst possible pain. A negative change (post surgery minus baseline) indicated an improvement. Percent change was calculated as: [(Month 24-Baseline)/Baseline]*100%.
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
percent change | -56.4 (92.5)

8. Secondary Outcome: Short Form 12 (SF-12v2) Physical Component Summary (PCS)
Description: The SF-12v2, comprising 12 questions related to health and wellbeing over the prior four weeks, was administered to subjects preoperatively and at all follow up visits. SF-12v2 represents overall subjective health status by measuring eight health-related parameters (each scored from 0 [poor health] to 100 [better health]): body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. First, the eight scales were standardized using means and standard deviations (SD) for the general US population. Second, PCS was scored by aggregating the eight scales using a standardized algorithm. Finally, PCS was standardized using a linear t-score transformation to have a mean of 50 and a SD of 10 in the general US population (expected range: 13-69).
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
units on a scale | 39.2 (8.0)

9. Secondary Outcome: Percent Change in Short Form 12 (SF-12v2) Physical Component Summary (PCS)
Description: The SF-12v2, comprising 12 questions related to health and wellbeing over the prior four weeks, was administered to subjects preoperatively and at all follow up visits. SF-12v2 represents overall subjective health status by measuring eight health-related parameters (each scored from 0 [poor health] to 100 [better health]): body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. First, the eight scales were standardized using means and standard deviations (SD) for the general US population. Second, PCS was scored by aggregating the eight scales using a standardized algorithm. Finally, PCS was standardized using a linear t-score transformation to have a mean of 50 and a SD of 10 in the general US population (expected range: 13-69). Percent change was calculated as [(Month 24 - Baseline)/Baseline]*100%.
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
percent change | 17.7 (31.4)

10. Secondary Outcome: Short Form 12 (SF-12v2) Mental Component Summary (MCS)
Description: The SF-12v2, comprising 12 questions related to health and wellbeing over the prior four weeks, was administered to subjects preoperatively and at all follow up visits. SF-12v2 represents overall subjective health status by measuring eight health-related parameters (each scored from 0 [poor health] to 100 [better health]): body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. First, the eight scales were standardized using means and standard deviations (SD) for the general US population. Second, MCS was scored by aggregating the eight scales using a standardized algorithm. Finally, MCS was standardized using a linear t-score transformation to have a mean of 50 and a SD of 10 in the general US population (expected range: 10-70).
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
units on a scale | 51.3 (7.9)

11. Secondary Outcome: Percent Change in Short Form 12 (SF-12v2) Mental Component Summary (MCS)
Description: The SF-12v2, comprising 12 questions related to health and wellbeing over the prior four weeks, was administered to subjects preoperatively and at all follow up visits. SF-12v2 represents overall subjective health status by measuring eight health-related parameters (each scored from 0 [poor health] to 100 [better health]): body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. First, the eight scales were standardized using means and standard deviations (SD) for the general US population. Second, MCS was scored by aggregating the eight scales using a standardized algorithm. Finally, MCS was standardized using a linear t-score transformation to have a mean of 50 and a SD of 10 in the general US population (expected range: 10-70). Percent change was calculated as [(Month 24 - Baseline)/Baseline]*100%.
Time Frame: Month 24
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | chronOS Strip
Number analyzed (Participants) | 55
percent change | 24.1 (29.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the Month 24 visit.
Arm/Group | chronOS Strip
Serious Adverse Events (participants affected / at risk) | 24/81
Other Adverse Events (participants affected / at risk) | 34/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | chronOS Strip (N=81)
Abnormal laboratory value (Blood and lymphatic system disorders) | 1
Cardiovascular (Cardiac disorders) | 6
Gastrointestinal (Gastrointestinal disorders) | 1
Surgery, other (Surgical and medical procedures) | 5
Infection, non-wound related (Infections and infestations) | 1
Dural tear (Injury, poisoning and procedural complications) | 2
Fever (Injury, poisoning and procedural complications) | 1
Cervical whiplash (Musculoskeletal and connective tissue disorders) | 1
Cervical disc rupture (Musculoskeletal and connective tissue disorders) | 1
Gout (Musculoskeletal and connective tissue disorders) | 1
Knee meniscus tear (Musculoskeletal and connective tissue disorders) | 1
Pain: back (Musculoskeletal and connective tissue disorders) | 2
Pain: back and legs (Musculoskeletal and connective tissue disorders) | 2
Surgery, index level (Surgical and medical procedures) | 3
Headache (Nervous system disorders) | 1
Neurological (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 2
Psychological (Psychiatric disorders) | 1
Genitourinary (Renal and urinary disorders) | 1
Routine vaginal delivery (Pregnancy, puerperium and perinatal conditions) | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Wound issues, other (Skin and subcutaneous tissue disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | chronOS Strip (N=81)
Neurological (Nervous system disorders) | 6
Pain, back (Musculoskeletal and connective tissue disorders) | 10
Pain, back and legs (Musculoskeletal and connective tissue disorders) | 11
Pain, legs (Musculoskeletal and connective tissue disorders) | 6
Pain, other (Musculoskeletal and connective tissue disorders) | 9

LIMITATIONS AND CAVEATS:
Limitations included lack of control arm, no hypothesis for primary endpoint, & qualitative sample size estimate. chronOS Strip was used according to its FDA-cleared labeling; other usage was outside the study scope and was not evaluated clinically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less